CLINICAL TRIAL: NCT05064787
Title: Evaluating the Feasibility of a Digital Health Coaching Program for Individuals Following CAR T Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pack Health (Industry)
Collaborators: M.D. Anderson Cancer Center (Other); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2021-0543
Record Dates: First submitted 2021-09-08; First posted 2021-10-01 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Lymphoma; Lymphoma, B-Cell; Leukemia; Multiple Myeloma; Mantle Cell Lymphoma; Follicular Lymphoma; Leukemia, Acute Lymphoblastic
Keywords: Receptors, chimeric antigen; Adult; hematologic neoplasms; digital health coaching
MeSH Terms: conditions — Lymphoma; Lymphoma, B-Cell; Leukemia; Multiple Myeloma; Lymphoma, Mantle-Cell; Lymphoma, Follicular; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Hematologic Neoplasms

STUDY DESIGN:
Intervention Model Description: A single cohort of 50 individuals receiving chimeric antigen receptor T cell therapy will be enrolled in the study, all of which will be enrolled in a 6-month digital health coaching program. Individuals will be enrolled from a single site, The University of Texas MD Anderson Cancer Center.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm Cohort Receiving Digital Health Coaching (Other): All study participants will be enrolled in a 6-month digital health coaching program.
  Interventions: Behavioral: Digital Health Coaching

INTERVENTIONS:
Behavioral: Digital Health Coaching — The digital health coaching program consists of weekly calls and delivery of evidence-based content across health and wellness domains (e.g. nutrition, exercise, physical, emotional and financial health) up to 4 times weekly via text, email or mobile application. The program is 6-months in duration and designed for engagement following CAR T cell infusion.

SUMMARY:
The aim of this study is to evaluate the feasibility of a digital health coaching program for, and to describe quality of life of, individuals in the 6 months following chimeric antigen receptor (CAR) T cell therapy. Up to 50 English-speaking individuals aged 18 and older who are to receive treatment with a CAR T cell therapy will be enrolled, all at The University of Texas MD Anderson Cancer Center. Participants must have internet access via smart phone, tablet, a computer, or another device with the capacity to receive calls, texts, or e-mails, as well as the electronic study assessments and will be excluded if they are unable to provide informed consent or have a prognosis of 6 months or less.

Consented participants will be enrolled in a 6-month digital health coaching program delivered via weekly calls from a Health Advisor coupled with the digital delivery of content. The program focuses on identification and escalation of treatment-related toxicity, communication with providers, and physical and psychosocial health following treatment. Health related quality of life (HRQoL) will be assessed with the Functional Assessment of Cancer Therapy-Lymphoma (FACT-L), health self-efficacy will be assessed by the Cancer Behavior Inventory-Brief (CBI-B), physical and mental health outcomes will be measured by the National Institutes of Health (NIH) Patient Reported Outcomes Measurement Information System (PROMIS) Global Health 10. Patient experience in managing CAR T specific care will be assessed with a 5-item questionnaire developed specifically for use in this study, focused on participants' confidence in understanding, identifying and managing symptoms, and communicating with providers. Study outcomes will contribute to knowledge about if and how a digital health intervention may be used to support individuals post-CAR T cell therapy.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 and older
* Able to read, speak and consent in English
* Confirmed treatment with any commercially available or investigational CAR T cell therapy.
* Internet access via smart phone, tablet, a computer, or another device with the capacity to receive calls, texts, or e-mails, as well as the electronic study assessments.
* Ability to engage in physical activity as evidenced by an Eastern Cooperative Oncology Group (ECOG) performance status score of less than or equal to 2

Exclusion Criteria:

* Individuals who are terminally ill, defined as individuals identified by their physician as likely having 6 months or less to live, or those individuals transitioned to comfort measures only (meaning only supportive care measures without curative focused treatment)
* Individuals for whom there is documentation of inability to provide consent in the medical record.
* Non-English speaking/reading individuals.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2022-03-11 (Actual); Primary Completion 2024-02-06 (Actual); Study Completion 2024-02-06 (Actual)

PRIMARY OUTCOMES:
Feasibility of the intervention | Through study completion, at month 6
  Feasibility is defined as a retention rate in the digital health coaching program greater than or equal to 60% at month 6
Acceptability | Through study completion, at month 6
  Acceptability will be assessed with a 3-item evaluation to address engagement, usefulness and relevance

SECONDARY OUTCOMES:
Cancer Behavior Inventory (CBI-B) | Enrollment, Months 1, 3, 6
  This 12-item instrument measures self-efficacy in coping with cancer across 7 domains. These include: Seeking and Understanding Medical Information, Emotion Regulation, Coping with Treatment Related Side Effects, Accepting Cancer/ Maintaining a Positive Attitude, Seeking Social Support, and Using Spiritual Coping. The instrument utilizes a 9-point response scale ranging from 1 "Not at all confident" to 9 "Confident".
Functional Assessment of Cancer Therapy-Lymphoma (FACT-Lym) | Enrollment, Months 1, 3, 6
  The FACT-lym is a 42-item assessment that measures self-reported quality of life across 4 domains: physical, functional, emotional and social and includes 15 additional items validated specifically for individuals with lymphoma. The instrument can be scored as a whole as well as within the individual domains.
National Institutes of Health (NIH) Patient Reported Outcomes Measurement Information System (PROMIS) Global Health 10 | Enrollment, Month 6
  Patient Reported Outcomes Measurement Information System (PROMIS) Global Health Scale is a ten item likert-scale survey that evaluates physical, social, and psychological well-being. The instrument consists of two scales, one for global physical health and one for global mental health.
Subjective Assessment of CAR T Management | Enrollment, Months 1, 3, 6
  a 5-item assessment of patients' experience in monitoring, managing, and reporting treatment related toxicities will be created specifically for use in this study and will mirror the response scale in the CBI-B. This includes a 9-point response scale ranging from 1 "Not at all confident" to 9 "Confident". The following items will be included: 1) Understand the treatment toxicities I may experience while receiving CAR T-cell therapy; 2) Identify the signs and symptoms of these toxicities; 3) Communicate symptoms to provider; 4) Manage symptoms according to provider's instructions; 5) Explain treatment to a healthcare provider.

OTHER OUTCOMES:
Socio-demographic, clinical, and treatment characteristics | Through study completion, at month 6
  Age, Race, Ethnicity, Sex at Birth, Gender Identity, Diagnosis, Treatment History, Co-morbid conditions
Health Care Utilization | Through study completion, at month 6
  ER visits and unplanned hospitalizations
Digital Engagement | Through study completion, at month 6
  Frequency, types and duration of engagement with the digital health coaching platform

CONTACTS AND LOCATIONS:
Overall Officials: Sherry Adkins, MSN, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas MD Anderson Cancer Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Beaupierre A, Kahle N, Lundberg R, Patterson A. Educating Multidisciplinary Care Teams, Patients, and Caregivers on CAR T-Cell Therapy. J Adv Pract Oncol. 2019 May-Jun;10(Suppl 3):29-40. doi: 10.6004/jadpro.2019.10.4.12. Epub 2019 May 1. PMID 33520344
- [Background] Buitrago J, Adkins S, Hawkins M, Iyamu K, Oort T. Adult Survivorship: Considerations Following CAR T-Cell Therapy. Clin J Oncol Nurs. 2019 Apr 1;23(2):42-48. doi: 10.1188/19.CJON.S1.42-48. PMID 30880816
- [Background] Chakraborty R, Sidana S, Shah GL, Scordo M, Hamilton BK, Majhail NS. Patient-Reported Outcomes with Chimeric Antigen Receptor T Cell Therapy: Challenges and Opportunities. Biol Blood Marrow Transplant. 2019 May;25(5):e155-e162. doi: 10.1016/j.bbmt.2018.11.025. Epub 2018 Nov 28. PMID 30500439
- [Background] Gajra A, Jeune-Smith Y, Kish J, Yeh TC, Hime S, Feinberg B. Perceptions of community hematologists/oncologists on barriers to chimeric antigen receptor T-cell therapy for the treatment of diffuse large B-cell lymphoma. Immunotherapy. 2020 Jul;12(10):725-732. doi: 10.2217/imt-2020-0118. Epub 2020 Jun 18. PMID 32552151
- [Background] Nabhan C, Jeune-Smith Y, Klinefelter P, Fillman J, Feinberg BA. Community Oncologists 'Perception and Adaptability to Emerging Chimeric Antigen T-Cell Therapy. J Clin Pathways. 2017;3(8):31-35.
- [Background] London S. Logistics of CAR T-cell therapy in real-world practice. The ASCO Post website ascopost.com/issues/may-25-2018/logistics-of-car-t-cell-therapy-in-real-world-practice Published May. 2018;25.
- [Background] Girault A, Ferrua M, Lalloue B, Sicotte C, Fourcade A, Yatim F, Hebert G, Di Palma M, Minvielle E. Internet-based technologies to improve cancer care coordination: current use and attitudes among cancer patients. Eur J Cancer. 2015 Mar;51(4):551-557. doi: 10.1016/j.ejca.2014.12.001. Epub 2015 Feb 4. PMID 25661828
- [Background] Madore S, Kilbourn K, Valverde P, Borrayo E, Raich P. Feasibility of a psychosocial and patient navigation intervention to improve access to treatment among underserved breast cancer patients. Support Care Cancer. 2014 Aug;22(8):2085-93. doi: 10.1007/s00520-014-2176-5. Epub 2014 Mar 18. PMID 24639035
- [Background] Green AC, Hayman LL, Cooley ME. Multiple health behavior change in adults with or at risk for cancer: a systematic review. Am J Health Behav. 2015 May;39(3):380-94. doi: 10.5993/AJHB.39.3.11. PMID 25741683
- [Background] Aapro M, Bossi P, Dasari A, Fallowfield L, Gascon P, Geller M, Jordan K, Kim J, Martin K, Porzig S. Digital health for optimal supportive care in oncology: benefits, limits, and future perspectives. Support Care Cancer. 2020 Oct;28(10):4589-4612. doi: 10.1007/s00520-020-05539-1. Epub 2020 Jun 12. PMID 32533435
- [Background] Heitzmann CA, Merluzzi TV, Jean-Pierre P, Roscoe JA, Kirsh KL, Passik SD. Assessing self-efficacy for coping with cancer: development and psychometric analysis of the brief version of the Cancer Behavior Inventory (CBI-B). Psychooncology. 2011 Mar;20(3):302-12. doi: 10.1002/pon.1735. PMID 20878830
- [Background] Hlubocky FJ, Webster K, Beaumont J, Cashy J, Paul D, Abernethy A, Syrjala KL, Von Roenn J, Cella D. A preliminary study of a health related quality of life assessment of priority symptoms in advanced lymphoma: the National Comprehensive Cancer Network-Functional Assessment of Cancer Therapy - Lymphoma Symptom Index. Leuk Lymphoma. 2013 Sep;54(9):1942-6. doi: 10.3109/10428194.2012.762977. Epub 2013 Feb 7. PMID 23320888
- [Background] Hays RD, Bjorner JB, Revicki DA, Spritzer KL, Cella D. Development of physical and mental health summary scores from the patient-reported outcomes measurement information system (PROMIS) global items. Qual Life Res. 2009 Sep;18(7):873-80. doi: 10.1007/s11136-009-9496-9. Epub 2009 Jun 19. PMID 19543809
- [Background] Neelapu SS. Managing the toxicities of CAR T-cell therapy. Hematol Oncol. 2019 Jun;37 Suppl 1:48-52. doi: 10.1002/hon.2595. PMID 31187535
- [Background] Amonoo HL, Kurukulasuriya C, Chilson K, Onstad L, Huffman JC, Lee SJ. Improving Quality of Life in Hematopoietic Stem Cell Transplantation Survivors Through a Positive Psychology Intervention. Biol Blood Marrow Transplant. 2020 Jun;26(6):1144-1153. doi: 10.1016/j.bbmt.2020.02.013. Epub 2020 Feb 20. PMID 32088365
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686